CLINICAL TRIAL: NCT04019704
Title: AXS-05-MDD-301: A Randomized, Double-Blind, Placebo-Controlled Trial of AXS-05 in Subjects With Major Depressive Disorder
Brief Title: A Trial of AXS-05 in Patients With Major Depressive Disorder
Acronym: GEMINI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AXS-05-MDD-301
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Depression; Major Depressive Disorder
Keywords: Depressive Disorder; Depressive Disorder, Major; Bupropion; Dextromethorphan; MDD; Dopamine Reuptake Inhibitor; AXS-05; NMDA Receptor Antagonist; Central Nervous System; CNS; Sigma-1 Receptor Agonist; Nicotinic Acetylcholine Receptor Antagonist; Norepinephrine Reuptake Inhibitor; Glutamate Modulator; Axsome Therapeutics; GEMINI; Serotonin Reuptake Inhibitor
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXS-05 (Experimental): AXS-05 (bupropion and dextromethorphan) oral tablets
  Interventions: Drug: AXS-05
- Placebo (Placebo Comparator): Placebo oral tablets to match AXS-05
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXS-05 — Oral AXS-05 tablets, taken daily for 6 weeks.
  Arms: AXS-05
Drug: Placebo — Placebo to match oral AXS-05 tablets, taken daily for 6 weeks.
  Arms: Placebo

SUMMARY:
A Phase 3, randomized, double-blind, placebo-controlled, multicenter trial of AXS-05 in patients with major depressive disorder (MDD).

DETAILED DESCRIPTION:
This study will evaluate AXS-05 in a randomized, double-blind, placebo-controlled study in patients with MDD. Eligible patients will be randomized in a 1:1 ratio to treatment with AXS-05 or placebo for 6 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 18 - 65
* Currently meets DSM-5 criteria for MDD
* Body Mass Index between 18 and 40 kg/m^2, inclusive

Key Exclusion Criteria:

* Suicide risk
* History of treatment resistance in current depressive episode
* History of electroconvulsive therapy, vagus nerve stimulation, transcranial magnetic stimulation or any experimental central nervous system treatment during the current episode or in the past 6 months
* Pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - Clinical Research Site, Phoenix, Arizona
  - Clinical Research Site, Little Rock, Arkansas
  - Clinical Research Site, Bellflower, California
  - Clinical Research Site, Beverly Hills, California
  - Clinical Research Site, Garden Grove, California
  - Clinical Research Site, Oakland, California
  - Clinical Research Site, Oceanside, California
  - Clinical Research Site, Panorama City, California
  - Clinical Research Site, Redlands, California
  - Clinical Research Site, Riverside, California
  - Clinical Research Site, San Diego, California
  - Clinical Research Site, Sherman Oaks, California
  - Clinical Research Site, Upland, California
  - Clinical Research Site, Coral Springs, Florida
  - Clinical Research Site, Hollywood, Florida
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Lauderhill, Florida
  - Clinical Research Site, North Miami, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Atlanta, Georgia
  - Clinical Research Site, Boise, Idaho
  - Clinical Research Site, Chicago, Illinois
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, Las Vegas, Nevada
  - Clinical Research Site, Berlin, New Jersey
  - Clinical Research Site, Cherry Hill, New Jersey
  - Clinical Research Site, Toms River, New Jersey
  - Clinical Research Site, Jamaica, New York
  - Clinical Research Site, Rochester, New York
  - Clinical Research Site, Staten Island, New York
  - Clinical Research Site, Hickory, North Carolina
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Middleburg Heights, Ohio
  - Clinical Research Site, Oklahoma City, Oklahoma
  - Clinical Research Site, Media, Pennsylvania
  - Clinical Research Site, Philadelphia, Pennsylvania
  - Clinical Research Site, Memphis, Tennessee
  - Clinical Research Site, Dallas, Texas
  - Clinical Research Site, Fort Worth, Texas
  - Clinical Research Site, Houston, Texas
  - Clinical Research Site, Wichita Falls, Texas
  - Clinical Research Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iosifescu DV, Jones A, O'Gorman C, Streicher C, Feliz S, Fava M, Tabuteau H. Efficacy and Safety of AXS-05 (Dextromethorphan-Bupropion) in Patients With Major Depressive Disorder: A Phase 3 Randomized Clinical Trial (GEMINI). J Clin Psychiatry. 2022 May 30;83(4):21m14345. doi: 10.4088/JCP.21m14345. PMID 35649167
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- See also: Axsome Therapeutics Website — http://www.axsome.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AXS-05 | Placebo
Started | 163 | 164
Completed | 123 | 147
Not Completed | 40 | 17

BASELINE CHARACTERISTICS:
Population: Participants randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | AXS-05 | Placebo | Total
Number analyzed (Participants) | 163 | 164 | 327
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (12.71) | 41.1 (13.78) | 41.6 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 117 | 215
  Male | 65 | 47 | 112
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 9 | 8 | 17
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 61 | 55 | 116
  White | 88 | 92 | 180
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in MADRS Total Score From Baseline to Week 6
Description: The primary objective of the study was to evaluate the efficacy of AXS-05 as measured by the Montgomery-Åsberg Depression Rating Scale (MADRS) for change in severity of depressive symptoms from baseline to Week 6. The MADRS is a 10-item scale and items are scored between 0-6 points. For each item, a score of 0 indicates the absence of symptoms, and a score of 6 indicates symptoms of maximum severity. A maximum total score is 60 points.
Time Frame: 6 weeks
Population: modified Intent-to-Treat (mITT) Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AXS-05 | Placebo
Number analyzed (Participants) | 156 | 162
score on a scale | 15.91 (0.921) | 12.04 (0.862)
Statistical Analysis 1: Comparison: AXS-05 vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were AEs with an onset date on or after the date of first dose. TEAEs were collected through 30 days after the last dose.
Description: Safety Population
Arm/Group | AXS-05 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/164
Serious Adverse Events (participants affected / at risk) | 1/162 | 0/164
Other Adverse Events (participants affected / at risk) | 100/162 | 74/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXS-05 (N=162) | Placebo (N=164)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Not related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXS-05 (N=162) | Placebo (N=164)
Dizziness (Nervous system disorders) | 26 (29) | 10 (12)
Nausea (Gastrointestinal disorders) | 21 (24) | 14 (14)
Headache (Nervous system disorders) | 13 (16) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 11 (11) | 5 (5)
Somnolence (Nervous system disorders) | 11 (11) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 9 (9) | 4 (4)
All Others, occurring in <5% of Subjects (General disorders) | 47 | 43 — All other events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT04019704/Prot_SAP_000.pdf